CLINICAL TRIAL: NCT02685631
Title: Radiation-Emitting SIR-Spheres in Non-resectable (RESIN) Liver Tumor Patient Study
Brief Title: Yttrium Y 90 Resin Microspheres Data Collection in Unresectable Liver Cancer: the RESIN Study
Acronym: RESiN
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel B. Brown, Principal Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICCGI1523; NCI-2015-01837 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC GI 1523 (Other: Vanderbilt University/Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2015-12-19; First posted 2016-02-19 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Localized Non-Resectable Adult Liver Carcinoma
Keywords: Hepatocellular carcinoma; Colorectal cancer; Neuroendocrine tumor; Cholangiocarcinoma; Breast cancer; Tumor of unknown primary; Pancreatic cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Neuroendocrine Tumors; Cholangiocarcinoma; Breast Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational/data registry collection: Patients receiving Yttrium-90 resin microspheres as part of care
  Interventions: Other: Yttrium-90 Resin Microspheres

INTERVENTIONS:
Other: Yttrium-90 Resin Microspheres — Data collection into the RESIN registry

SUMMARY:
This research registry studies Yttrium Y 90 resin microspheres in collecting data from patients with liver cancer not capable of being removed by surgery (unresectable) for the radiation-emitting Selective Internal Radiation-Spheres (SIR-spheres) in non-resectable (RESIN) liver tumor registry. The information generated will help doctors better understand treatment patterns involving Y90 therapy, gain additional insights in the long-term outcomes for patients, as well as guide future research for using Y90 therapy, especially for those conditions where data is currently very limited or lacking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The principal objective of the RESIN registry is to evaluate response to therapy using objective response criteria such as modified Response Evaluation Criteria in Solid Tumors (mRECIST) or European Association for Study of the Liver (EASL). The response criteria used will depend on tumor type treated and local policies as this is a registry and not a formal research study. Secondary criteria include overall survival, time to progression (TTP) and toxicity.

OUTLINE:

Patients receiving Yttrium Y90 resin microspheres treatment as part of their overall oncologic management are added in the RESIN registry database to collect and document information including: patient demographics (gender/age), previous oncologic treatments, details of Yttrium Y90 resin microspheres treatment, and to track outcomes and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving SIR-Spheres therapy to the liver for the first time.
* Provision of written informed consent.
* Age 18 and older.

Exclusion Criteria:

1. Prior completion of Y90 therapy to the liver (SIR-Spheres, TheraSpheres, or any other liver-targeted therapy involving the use of radiation-emitting spheres).

   -Patients who have received Y90 treatment in the past and who are returning for another Y90 treatment are ineligible, even if new areas are being targeted.
2. Need for surrogate consent. Patients unable to consent on their own behalves are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary and secondary liver cancer receiving SIR Spheres® microspheres (Y90 resin microspheres) treatment as part of their overall oncologic management
Sampling Method: Non-Probability Sample
Enrollment: 1653 (Actual)
Dates: Start 2015-07; Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Response to treatment with Y90 microspheres either as mono therapy or as part of multidisciplinary management of their specific disease | Up to 1 year after the first treatment
  Response to treatment is the initial measure of treatment efficacy. This can be measured using objective criteria such as the modified Response Evaluation Criteria in Solid Tumors (mRECIST) or European Association for Study of Liver Cancer (EASL) criteria depending on local policy and tumor type.

SECONDARY OUTCOMES:
Treatment related toxicity assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v4) measures | Up to 1 year after the first treatment
  Overall toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v4) measures. Tracking this outcome can help define optimal combinations of Y90 plus systemic or biologic therapy to be used in formal research studies in the future
Overall Survival | 2 years
  As noted above, overall survival is the optimal outcome measure with any oncologic therapy. However, the majority of patients will receive additional therapy after progressing on a given treatment regimen. For this reason, overall survival assessment with Y90 is a secondary, rather than a primary assessment endpoint in this registry study.
Time to Progression | 2 years
  Overall survival is the definitive measure of any oncologic therapy. However, many if not all patients receive other treatments at the time of tumor progression. For this reason TTP may be the most accurate measure of oncologic efficacy following Y90 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Brown, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (42):
- United States (42):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona Health Sciences, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Denver, Colorado
  - Sky Ridge Medical Center, Englewood, Colorado
  - Christiana Care Health System, Wilmington, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - Baptist Hospital of Miami, Miami, Florida
  - University of Miami, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cancer Treatment Centers of America, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health- Lenox Hill Hospital, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Methodist Health System, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Utah, Salt Lake City, Utah
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided
We plan on reporting group outcomes by tumor type or subtype. Individual records will be subject to HIPAA rules

REFERENCES:
- [Derived] Zhou W, Du L, Brown DB, Shah RP, Sze DY. Outcomes Analysis of Yttrium-90 Radioembolization for Tumors Other Than Metastatic Colorectal Cancer from the Radiation-Emitting SIR-Spheres in Nonresectable (RESiN) Registry. J Vasc Interv Radiol. 2024 Nov;35(11):1591-1600.e3. doi: 10.1016/j.jvir.2024.07.006. Epub 2024 Jul 14. PMID 39009301
- [Derived] Emmons EC, Bishay S, Du L, Krebs H, Gandhi RT, Collins ZS, O'Hara R, Akhter NM, Wang EA, Grilli C, Brower JS, Peck SR, Petroziello M, Abdel Aal AK, Golzarian J, Kennedy AS, Matsuoka L, Sze DY, Brown DB. Survival and Toxicities after 90Y Transarterial Radioembolization of Metastatic Colorectal Cancer in the RESIN Registry. Radiology. 2022 Oct;305(1):228-236. doi: 10.1148/radiol.220387. Epub 2022 Jun 28. PMID 35762890
- [Derived] Wong TY, Zhang KS, Gandhi RT, Collins ZS, O'Hara R, Wang EA, Vaheesan K, Matsuoka L, Sze DY, Kennedy AS, Brown DB. Long-term outcomes following 90Y Radioembolization of neuroendocrine liver metastases: evaluation of the radiation-emitting SIR-spheres in non-resectable liver tumor (RESiN) registry. BMC Cancer. 2022 Mar 1;22(1):224. doi: 10.1186/s12885-022-09302-z. PMID 35232410
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/